CLINICAL TRIAL: NCT06810297
Title: Effect of a Therapeutic Exercise and an Education Program on Sexual Function and Experience in People With Endometriosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Laura Fuentes Aparicio, Assistant Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SEX-ENDOMETRIO-UV
Record Dates: First submitted 2025-01-14; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis; Sexual Function; Sex Behavior
Keywords: Endometriosis; Sexual Function; Sexual Experience
MeSH Terms: conditions — Endometriosis; Sexual Behavior | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Exercise (Active Comparator): They will recive the therapeutic exercise program.
  Interventions: Procedure: Therapeutic Exercise
- Therapeutic exercise and sexual education (Experimental): They will receive ta combined program, which will combine therapeutic exercise with a sexual education classes.
  Interventions: Combination Product: Therapeutic exercise and sexual education

INTERVENTIONS:
Procedure: Therapeutic Exercise — It will consist of an 8-week intervention divided into 2 weekly sessions, in which functional exercise will be combined with aerobic exercise. A progressive protocol will be carried out.The sessions will last approximately 60 minutes divided into a first aerobic part which will serve as a warm-up for the functional part, then a main part with approximately 6 exercises and, finally, a cool-down of 3 to 5 minutes with relaxation exercises and stretching.
  Arms: Therapeutic Exercise
Combination Product: Therapeutic exercise and sexual education — The sexual education part will consist of a 4-week intervention divided into 1 session every two weeks in an online format, in which topics related to the pathology and self-knowledge will be addressed. The sessions will last approximately 60 minutes, divided into a first part of reception and welcome of the group (lasting approximately 5-10 minutes), then the main content will be divided differently in each session (the explicit content of each session will be detailed later) and will end with a farewell and closing of the online session (lasting approximately 5-10 minutes) together with the explanation of the homework.
  In addition, they will also carry out the therapeutic exercise protocol.
  Arms: Therapeutic exercise and sexual education

SUMMARY:
This is a randomized clinical trial that will be carried out in people with endometriosis divided into two groups: the experimental group (EG) that will receive therapeutic exercise combine with sexual education, and the control group (CG) who will receive the therapeutic exercise program.

The participants will be evaluated at three moments: before starting the study (T1), after the 8-week treatment program (T2) and after 4 weeks of follow-up in which they will be encouraged to continue with the treatment (T3). Objective and subjective data of the participants will be evaluated. T1 will be assessed with a sociodemographic questionnaire and the FSFI and MSSCQ surveys. T2 and T3 will assess blood pressure, heart rate, variability of the autonomic system, the ability to dissociate the lumbopelvic movement from the thoracolumbar, measurement of the muscles of the transverse, internal and external obliques, the distance between the rectus abdominis and the pelvic floor, subjective perception of effort during exercise and subjective perception of orgasmic intensity.

ELIGIBILITY:
Inclusion Criteria:

* People of legal age (over 18 years old)
* Not older than 50 years old
* Currently residing in Spain
* Spanish speakers
* With a medical diagnosis of endometriosis
* Without any other associated gynecological pathology

Exclusion Criteria:

* Minors
* People over 50 years old
* Those with cognitive limitations that prevent them from completing the different questionnaires used
* People who are involved in litigation processes
* People with gynecological pathologies other than endometriosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Quality of Life - Sexual Function | Measurements will be taken prior to the intervention (week 0 of the program), after the intervention has ended (week 8 of the program) and one month after the intervention has ended (week 12 of the program).
  The Index of Female Sexual Function (IFSF) will be used. It is a multidimensional self-reported instrument for the evaluation of female sexual function.
  The scores for the same domain are added together and multiplied by the factor that corresponds to each domain. The total score is obtained by adding the scores for the 6 domains. A score of 0 in any of the domains indicates a lack of sexual activity in the last month.The maximum total score will be 36 points and the minimum 2. The higher the score, the better the sexual function.
Quality of Life - Sexual self-concept | Measurements will be taken prior to the intervention (week 0 of the program), after the intervention has ended (week 8 of the program) and one month after the intervention has ended (week 12 of the program).
  Multidimensional Scale of Sexual Concept (MSSCQ) will be used. It is a multidimensional self-reported instrument for the evaluation of sexual self- concept.
  Each answer has a score of 0 to 4 points. The higher the score, the better the sexual assertiveness and sexual self-concept. There are a total of 16 questions. The maximum score is 64 points and the minimum is 0.

SECONDARY OUTCOMES:
Quality of Life - Pleasure | Measurements will be taken prior to the intervention (week 0 of the program), after the intervention has ended (week 8 of the program) and one month after the intervention has ended (week 12 of the program).
  Visual Analogue Scale (VAS) of pleasure will be used. Orgasmic intensity is reported through a Likert scale (0-10) and a chromatic gradation, which fluctuate from 0 (white), corresponding to the absence of orgasmic intensity, to 10 (deep red), corresponding to the highest level of orgasmic intensity.
Physical-Funcionality - Motor control | Measurements will be taken prior to the intervention (week 0 of the program), after the intervention has ended (week 8 of the program) and one month after the intervention has ended (week 12 of the program).
  Determine motor control: clinical test of lumpopelvic and thoracolumbar dissociation will be used.
  The clinical test assesses the ability to dissociate lumbopelvic movement from that of the thoracolumbar junction, and to evaluate the inter-rater reliability of the test in individuals with and without low back pain (LBP) when performed by experienced and novice therapists. A clinical scale was developed to characterise quality of performance of lumbopelvic motion with limited motion at the thoracolumbar junction. The patient is asked to flex the trunk to see if there is lumbopelvic dissociation.
Physical-Funcionality- Pelvic floor and abdominal ultrasound | Measurements will be taken prior to the intervention (week 0 of the program), after the intervention has ended (week 8 of the program) and one month after the intervention has ended (week 12 of the program).
  The ultrasound will measure muscle tone. This tone will be assessed in different situations. Measurement of basal tone, tone at maximum contraction, tone at Valsalva and tone at cough.

OTHER OUTCOMES:
Excitation | Measurements will be taken prior to the intervention (week 0 of the program), after the intervention has ended (week 8 of the program) and one month after the intervention has ended (week 12 of the program).
  Sphygmomanometer will be used to measure the patients' arousal. Blood pressure will be measured to assess the level of arousal. Blood pressure is controlled by the autonomic system, which is also responsible for arousal. The higher the blood pressure, the greater the activation of the sympathetic system. Lower blood pressures indicate that the parasympathetic system is more active.
Excitation | Measurements will be taken prior to the intervention (week 0 of the program), after the intervention has ended (week 8 of the program) and one month after the intervention has ended (week 12 of the program).
  Electrocardiogram will be used to measure the patients' arousal. The electrocardiogram measures heart rate. It is also measured by the autonomic nervous system, so it is closely related to excitement. During excitement, a person's heart rate increases.
Excitation | Measurements will be taken prior to the intervention (week 0 of the program), after the intervention has ended (week 8 of the program) and one month after the intervention has ended (week 12 of the program).
  eSense skin response will be used to measure the patients' arousal. The activation of the sympathetic and parasympathetic systems is recorded through the skin. Higher values and the red colour measured with the eSense device indicate that the sympathetic system is more active. If the values tend to 0 and the colour is green, there is more activation of the parasympathetic system.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Laura Fuentes Aparicio, Valencia
  - University of Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No